CLINICAL TRIAL: NCT03211533
Title: CareToy Observational Study: Early Identification of Infants at Risk of Cerebral Palsy
Brief Title: Early Identification of Infants at Risk of Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: IRCCS Fondazione Stella Maris (Other)
Responsible Party: Sponsor
Other Study IDs: RF-2013-02358095
Record Dates: First submitted 2017-06-28; First posted 2017-07-07 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2019-10

CONDITIONS: Cerebral Palsy; Preterm Infant
Keywords: infants at risk of cerebral palsy; MRI; general movements
MeSH Terms: conditions — Cerebral Palsy; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This observational study aims to early identify, through a rigorous and standardized follow-up, infants at high risk for Cerebral Palsy. After the consent agreement firmed by the parents, infants born at term or preterm with ultrasonographic evidence of brain injury considered at risk for neurodevelopmental disorders will be strictly monitored during the first months of life performing a periodic neurological assessment (Prechtl's General Movement (GMA) and the Hammersmith Infant Neurological Examination) at term age and around 3 months of post term age. Moreover, to study more accurately the brain injury early identified by ultrasonographic brain exam, around 6 weeks of post-term age the enrolled infants will perform, as recommended in infants at risk, brain Magnetic Resonance (RM).

Thanks to the high predictability power of the combination of the clinical observation with the neuroimaging infants at high risk of CP will be early detect. Selected infants, considered at high risk for CP will have the opportunity to perform an home based and family centered early intervention later than 3 post term age.

DETAILED DESCRIPTION:
Scientific literature review shows evidence that early intervention, especially when performed in the first months of life, when the brain plasticity shows its great expressivity, has positive effects on neurodevelopmental outcomes. In this framework the early identification of infants at risk for neurodevelopmental disorders is a major prerequisite to start very early an intervention programme. To families of infants, born in Neonatal Units involved in this study, will be asked with written informed consent, to participate in this observational study that aims to early identify, through a rigorous and standardized follow-up, infants at high risk for CP. Infants born at term or preterm with ultrasonographic evidence of brain injury considered at risk for neurodevelopmental disorders will be strictly monitored during the first months of development by the clinical team (Child Neurologists and Neonatologists) performing a periodic neurological assessment through examination of the Prechtl's General Movement (GMA) and the Hammersmith Infant Neurological Examination, at term age and around 3 months of post term age. Moreover, to study more accurately the brain injury early identified by ultrasonographic brain exam, within 6 weeks post-term age enrolled infants will perform, as recommended in infants at risk, brain Magnetic Resonance (RM). During the conventional RM examination, when possible, a fMRI perceptive task will be also performed to evaluate possible predictor factors to the responsiveness to the early intervention.

Thanks to the high predictability power of the combination of the clinical observation with the neuroimaging infants at high risk of CP will be early detect. Selected infants, considered at high risk for CP will have the opportunity to perform an home based and family centered early intervention later than 3 post term age.

ELIGIBILITY:
Inclusion Criteria:

* neurological signs (Hammersmith Infant Neurological Examination/General Movement Assessment according Precthl's).
* signs of brain injury identified at ultrasound brain exam

Exclusion Criteria:

* brain malformations
* severe sensory deficits

Max Age: 5 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: For this observational study will be enrolled infants, born a term or preterm, with very early neurological signs (at term age) and evidences of brain lesion during ultrasound brain screening that are considered at risk for the development of CP.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-07-22 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-23 (Actual)

PRIMARY OUTCOMES:
Fidgety Movements at 12 weeks (post-term age) | 12 weeks post-term age
  The Prechtl's General Movements Assessment is a non-invasive and cost-effective way to identify neurological issues which may lead to cerebral palsy and other developmental disabilities. The Fidgety movements are usually assessed between 9-20 weeks post-term age, showing the best expression at 12 weeks post term age. Infants whose Fidgety movements are absent or abnormal are at higher risk of neurological conditions, in particular for cerebral palsy.

SECONDARY OUTCOMES:
Writhing Movements at 40 weeks (term age) | 40 weeks (term age)
  The 'writhing movements' (described in the Prechtl's General Movements Assessment) are present from term age until 8 weeks post-term age. The evaluation at 40 weeks is a key point for the assessment both in preterm and at term infants. Infants whose writhing movements are abnormal could be considered at risk for neurodevelopmental disabilities; they have been carefully monitored in the fidgety period (see primary outcome measure).
Magnetic resonance imaging rating scale | up to 6 weeks (post-term age)
  Infants recruited will perform, according to gold standard clinical guidelines, a MRI study of the brain lesion previously identified with brain ultrasound. MRI will allow to better study the type of lesion. It will be quantified according to a validated visual semi-quantitative rating scale that uses a reliable and valid anatomical template for a graphical representation of abnormal MRI findings with detailed scoring of relative brain structures. During the MRI a task of fMRI will be performed to identify predictors of response to treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Stella Maris, Calambrone, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Franchi De' Cavalieri M, Filogna S, Martini G, Beani E, Maselli M, Cianchetti M, Dubbini N, Cioni G, Sgandurra G; CareToy-R Consortium. Wearable accelerometers for measuring and monitoring the motor behaviour of infants with brain damage during CareToy-Revised training. J Neuroeng Rehabil. 2023 May 6;20(1):62. doi: 10.1186/s12984-023-01182-z. PMID 37149595
- [Derived] Menici V, Antonelli C, Beani E, Mattiola A, Giampietri M, Martini G, Rizzi R, Cecchi A, Cioni ML, Cioni G, Sgandurra G; Caretoy-R Consortium. Feasibility of Early Intervention Through Home-Based and Parent-Delivered Infant Massage in Infants at High Risk for Cerebral Palsy. Front Pediatr. 2021 Jul 19;9:673956. doi: 10.3389/fped.2021.673956. eCollection 2021. PMID 34350144
- [Derived] Sgandurra G, Beani E, Giampietri M, Rizzi R, Cioni G; CareToy-R Consortium. Early intervention at home in infants with congenital brain lesion with CareToy revised: a RCT protocol. BMC Pediatr. 2018 Sep 5;18(1):295. doi: 10.1186/s12887-018-1264-y. PMID 30185165